CLINICAL TRIAL: NCT01064635
Title: Letrozole Adjuvant Therapy Duration (LEAD) Study: Standard Versus Long Treatment. A Phase III Trial in Post-Menopausal Women With Early Breast Cancer.
Brief Title: Letrozole in Treating Breast Cancer in Postmenopausal Women With Stage I, II, or III Breast Cancer Previously Treated With Tamoxifen (GIM4)
Acronym: GIM4
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Lucia Del Mastro,MD, Principal Invesitagator, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000665188; GIM-4-LEAD (Other: Consorzio oncotech); 2005-001212-44 (EudraCT Number); EU-21003
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

ARMS (2):
- Letrozole for 3-2 years (Active Comparator): Patients pre-treated with TAM for 2-3 years will receive letrozole 2,5 mg/die for 3-2 years. Total duration of early adjuvant endocrine therapy: 5 years
  Interventions: Drug: Letrozole
- Letrozole for 5 year (Experimental): Patients pre-treated with TAM for 2-3 years will receive letrozole 2,5 mg/die for additional 5 years. Total duration of early adjuvant endocrine therapy: 7 years for patients pretreated with 2 years of TAM and 8 years for patients pre-treated with 3 years of TAM
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — letrozole for 2-3 years after Tam
  Arms: Letrozole for 3-2 years
Drug: Letrozole — Letrozole for 5 years after Tam
  Arms: Letrozole for 5 year

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Letrozole may fight breast cancer by lowering the amount of estrogen the body makes. It is not yet known which regimen of letrozole is most effective in treating breast cancer in postmenopausal women who have received tamoxifen.

PURPOSE: This randomized phase III trial is comparing different regimens of letrozole to see how well they work in treating postmenopausal women with stage I, stage II, or stage III breast cancer previously treated with tamoxifen.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the disease-free survival of previously treated, post-menopausal women with early-stage breast cancer treated with standard- (2-3 years of tamoxifen followed by 2-3 years of letrozole) versus long-treatment (2-3 years of tamoxifen followed by 5 years of letrozole) adjuvant letrozole.

Secondary

* To compare the overall survival of these patients.
* To compare the safety of these patients.

OUTLINE: Patients are randomized to 1 or 2 treatment arms.

* Arm I (standard treatment): Patients previously treated with tamoxifen for 2 years receive letrozole for an additional 3 years; patients previously treated with tamoxifen for 3 years receive letrozole for an additional 2 years; and patients previously treated with tamoxifen for 2-3 years receive letrozole , so the total duration of the endocrine treatment (i.e., tamoxifen followed by letrozole) is 5 years.
* Arm II (long treatment): Patients receive letrozole for an additional 5 years regardless of the duration of the previous tamoxifen treatment.

ELIGIBILITY:
INCLUSION CRITERIA

* Signed informed consent prior to beginning protocol specific procedures.
* Histologically proven breast cancer at the first diagnosis with tumor stage I-II-III. Patients with histologically documented (microscopic) infiltration of the skin (pT4) will also be eligible.
* Axillary Nodal status allowed: Nx, pNo, pN1, pN2, pN3.
* Postmenopausal status defined by one of the following:

  * Age > 55 years with cessation of menses
  * Age < 55 years but not spontaneous menses for at least 1 year
  * Age < 55 years and spontaneous menses within the past 1 year, but currently amenorrheic (e.g. spontaneous, or secondary to hysterectomy), AND with postmenopausal gonadotrophin levels (luteinizing hormone and follicle stimulating hormone levels >40 IU/L) or postmenopausal estradiol levels (<5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved.
  * Bilateral oophorectomy
* Adjuvant TAM received for at least 2 years and not more than 3 years and 3 months. Patients treated with adjuvant chemotherapy, are required to have begun receiving TAM within 3 months after the completion of chemotherapy.
* Definitive surgical treatment must be either mastectomy or breast conserving surgery, with axillary lymph node dissection or sentinel node biopsy for operable breast cancer.
* ECOG/WHO performance Status 0-1. Patients must be accessible for treatment and follow-up.
* Concomitant treatment with biphosphonates are allowed and should be recorded during the trial.

EXCLUSION CRITERIA

* Male patients.
* Any locally advanced (T4) or inflammatory breast cancer. However, patients with microscopic infiltration of the skin (pT4) will be eligible.
* Patients with distant metastases. Any suspicious manifestation requires appropriate investigation to exclude metastases.
* Histology other than adenocarcinoma.
* Patients with previous or concomitant (not breast cancer) malignancy within the past 5 years EXCEPT adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix. Patients who have had a previous other malignancy must have been disease free for 5 years.
* Patients with other non-malignant systemic diseases (cardiovascular, renal, hepatic, lung embolism, etc.) which would prevent prolonged follow-up.
* Use of hormone Replacement Therapy within four weeks before randomization.
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational regimen within 30 days prior to study entry.
* Concurrent treatment with any other anti-cancer therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2056 (Actual)
Dates: Start 2005-08; Primary Completion 2015-08 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 6 years after the last patient enters the study

SECONDARY OUTCOMES:
Overall survival | 6 years after the last patient enters the study
Safety | 6 years after the last patient enters the study

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Del Mastro, MD, Principal Investigator — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Locations (1):
- Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy

REFERENCES:
- [Derived] Del Mastro L, Mansutti M, Bisagni G, Ponzone R, Durando A, Amaducci L, Campadelli E, Cognetti F, Frassoldati A, Michelotti A, Mura S, Urracci Y, Sanna G, Gori S, De Placido S, Garrone O, Fabi A, Barone C, Tamberi S, Bighin C, Puglisi F, Moretti G, Arpino G, Ballestrero A, Poggio F, Lambertini M, Montemurro F, Bruzzi P; Gruppo Italiano Mammella investigators. Extended therapy with letrozole as adjuvant treatment of postmenopausal patients with early-stage breast cancer: a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2021 Oct;22(10):1458-1467. doi: 10.1016/S1470-2045(21)00352-1. Epub 2021 Sep 17. PMID 34543613
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT01064635